CLINICAL TRIAL: NCT04364763
Title: A Phase 2, Randomized, Placebo-Controlled Study to Evaluate the Effect of RBT-9 on Progression of COVID-19 in High-Risk Individuals (The PREVENT Study)
Brief Title: A Study to Evaluate the Effect of RBT-9 on Progression of COVID-19 in High-Risk Individuals (The PREVENT Study)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Enrollment feasibility
Sponsor: Renibus Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REN-005
Record Dates: First submitted 2020-04-20; First posted 2020-04-28 (Actual); Results first posted 2023-03-29 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — tin protoporphyrin IX; Sodium Chloride; Saline Solution

STUDY DESIGN:
Intervention Model Description: 2:1 randomization to receive RBT-9:Placebo
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- RBT-9 (90 mg) (Experimental): RBT-9 (90mg) will be administered intravenously over a 120-minute period on Day 1.
  Interventions: Drug: RBT-9 (90 mg)
- Placebo (Placebo Comparator): 0.9% sodium chloride (normal saline) will be administered intravenously over a 120-minute period on Day 1.
  Interventions: Drug: 0.9% sodium chloride (normal saline)

INTERVENTIONS:
Drug: RBT-9 (90 mg) — Subjects will receive a single dose and study duration will be approximately 60 days per subject.
  Arms: RBT-9 (90 mg)
Drug: 0.9% sodium chloride (normal saline) — Subjects will receive a single dose and study duration will be approximately 60 days per subject.
  Arms: Placebo

SUMMARY:
The overall objective is to evaluate the efficacy, tolerability, and safety of a single dose of RBT-9 versus placebo in coronavirus disease 2019 (COVID-19) infection in non-critically ill adults who are at high risk of progression.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, ≥18 years of age at Screening.
2. Confirmed infection with SARS-CoV-2.
3. High risk of COVID-19 disease progression, defined as:

   1. 18-69 years of age with lymphopenia AND 1 additional risk factor (described below)
   2. 18-69 years of age without lymphopenia AND 2 risk factors (described below)
   3. ≥70 years of age with lymphopenia OR 1 other risk factor (described below)

   Risk Factors:
   * Documented history of coronary artery disease
   * Heart failure (New York Heart Association Class 3 or 4)
   * Chronic lung disease (eg, asthma or chronic obstructive pulmonary disease) requiring treatment
   * Documented history of stroke
   * Diabetes mellitus, requiring at least 1 prescription medicine for management
   * Documented chronic kidney disease with an estimated glomerular filtration rate <30 mL/min, not on dialysis
   * Obesity (Class 2 or 3; body mass index >34.9 kg/m2)
   * On immunosuppressive therapy
   * Oxygen saturation between 90 and 95% with or without supplemental oxygen
4. Admitted to a hospital for observation and/or treatment (controlled facility may include an emergency room, urgent care facility, temporary/modular hospital, infusion center, clinical research unit, etc).
5. If female, must be postmenopausal, surgically sterile, or if of childbearing potential, must be practicing 2 effective methods of birth control during the study and through 30 days after completion of the study.
6. For females of childbearing potential, a urine pregnancy test must be negative at the Screening Visit.
7. If male, must be surgically sterile or willing to practice 2 effective methods of birth control during the study and through 30 days after completion of the study.
8. Must be willing and able to give informed consent and comply with all study procedures.

Exclusion Criteria:

1. Anticipated need for ICU care and/or ventilatory support (invasive or noninvasive) within 24 hours.
2. Evidence of acute cardiac injury, as determined by the Investigator at the time of Screening. This may be based upon clinical signs and symptoms, ECG findings, or elevated troponin I levels.
3. Evidence of acute kidney injury not due to pre-renal azotemia or urinary tract obstruction at the time of Screening.
4. Oxygen saturation <90% on supplemental oxygen with a nasal cannula, including high-flow oxygen at the time of Screening.
5. Requires non-invasive ventilation at the time of Screening.
6. Requires dialysis at the time of Screening.
7. Has received or is receiving anti-IL-6 therapies (eg, Tocilizumab, Sarilumab, Siltuximab, etc) for the treatment of COVID-19; subjects receiving anti-IL-6 therapies for underlying medical conditions unrelated to COVID-19 are not excluded from eligibility.
8. Pregnant or lactating.
9. History of photosensitivity or active skin disease that, in the opinion of the Investigator, could be worsened by RBT-9.
10. Known hypersensitivity or previous anaphylaxis to RBT-9 (stannous protoporphyrin) or any tin-based product.
11. Treatment with an investigational drug or participation in an interventional trial within 30 days prior to the first dose of study drug.
12. Inability to comply with the requirements of the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2020-08-05 (Actual); Primary Completion 2021-09-02 (Actual); Study Completion 2021-09-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - New Smyrna Beach, FL, New Smyrna Beach, Florida
  - Berkley, MI, Berkley, Michigan
  - El Paso, TX, El Paso, Texas
  - Fort Worth, TX, Fort Worth, Texas
  - Houston, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | RBT-9 (90 mg) | Placebo
Started | 28 | 14
Completed (Day 56 Study Visit) | 26 | 12
Not Completed | 2 | 2
Not completed — Death | 1 | 2
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RBT-9 (90 mg) | Placebo | Total
Number analyzed (Participants) | 28 | 14 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 7 | 27
  >=65 years | 8 | 7 | 15
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.6 (16.59) | 57.6 (17.11) | 55 (16.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 9 | 26
  Male | 11 | 5 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 2 | 17
  Not Hispanic or Latino | 13 | 12 | 25
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 5 | 7
  White | 21 | 6 | 27
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 2 | 7
Region of Enrollment [Number; unit: participants]
  United States | 28 | 14 | 42

OUTCOME MEASURES:

1. Primary Outcome: Evaluate the Effect of RBT-9 Versus Placebo on Clinical Status of COVID-19 Patients as Measured Using the 8-point World Health Organization (WHO) Ordinal Clinical Scale
Description: Determining severity of COVID-19 in patients measured using the 8-point World Health Organization (WHO) Ordinal Clinical Scale which measures the clinical status of a subject at the first assessment of a given day with category 1, most favorable, and category 8, least favorable (1. Ambulatory, no limitation of activities; 2. Ambulatory, limitation of activities; 3. Hospitalized, no oxygen therapy; 4. Hospitalized, oxygen by mask or nasal prongs; 5. Hospitalized, non-invasive ventilation or high-flow oxygen; 6. Hospitalized, intubation and mechanical ventilation; 7. Hospitalized, ventilation plus additional organ support - pressors, renal replacement therapy [RRT], extracorporeal membrane oxygenation [ECMO]; 8. Death)
Time Frame: baseline and 7 days, baseline and 28 days
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | RBT-9 (90 mg) | Placebo
Number analyzed (Participants) | 28 | 14
units on a scale
  Day 7 | -1.0 [-1.6 to -0.5] | -0.0 [-0.8 to 0.8]
  Day 28 | -1.2 [-1.8 to -0.7] | -0.6 [-1.5 to 0.4]
Statistical Analysis 1: Comparison: RBT-9 (90 mg) vs Placebo; Test type: Superiority; p = 0.0352, Mixed Models Analysis — p-value is for Day 7
Statistical Analysis 2: Comparison: RBT-9 (90 mg) vs Placebo; Comparison made for Day 7 and Day 28; Test type: Superiority; p = 0.2350, Mixed Models Analysis — p-value is for Day 28

ADVERSE EVENTS:
Time Frame: Subjects will receive a single dose of RBT-9 or placebo and study duration will be approximately 56 +/- 4 days per subject.
Description: AEs and SAEs determined to be related to COVID-19 were not reportable under the requirements of this protocol. Rather, they were reported as complications or signs/symptoms of COVID.
Arm/Group | RBT-9 (90 mg) | Placebo
All-Cause Mortality (participants affected / at risk) | 1/28 | 2/14
Serious Adverse Events (participants affected / at risk) | 3/28 | 1/14
Other Adverse Events (participants affected / at risk) | 6/28 | 4/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RBT-9 (90 mg) (N=28) | Placebo (N=14)
Myocardial Infarction (Cardiac disorders) | 0 (0) | 1 (1) — Myocardial infarction resulting in death
Cerebral Infarct (Nervous system disorders) | 1 (1) | 0 (0) — Acute right posterior cerebral infarct
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Pneumonia
Lung mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Left lung mass
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | RBT-9 (90 mg) (N=28) | Placebo (N=14)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1)
Onychomycosis (Infections and infestations) | 0 (0) | 1 (1)
Tinea cruris (Infections and infestations) | 0 (0) | 1 (1)
Paresthesia (Nervous system disorders) | 2/2 (2) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-15): https://cdn.clinicaltrials.gov/large-docs/63/NCT04364763/Prot_SAP_001.pdf